CLINICAL TRIAL: NCT06683443
Title: Assessing the Effects of Robotic Pets on Patients With Dementia in the Acute Care Hospital Setting
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Sarasota Memorial Health Care System (Other)
Responsible Party: Principal Investigator, Joanna D'Elia, Adv Specialty Program Coord, Clinical Specialty Programs, Sarasota Memorial Health Care System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 23-MEDI-96
Record Dates: First submitted 2024-07-19; First posted 2024-11-12 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Dementia; Delirium
Keywords: dementia; memory impairment; delirium
MeSH Terms: conditions — Dementia; Delirium; Memory Disorders

STUDY DESIGN:
Intervention Model Description: A total of 106 patients, ages 65 years or older, with dementia who are admitted to the designated medical-surgical units at SMHCS will be enrolled in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robotic Pet (Experimental): The intervention group will receive the robotic Joy for All™ pet.
  Interventions: Behavioral: Robotic Joy for All™ pet
- Control (No Intervention): Control group will receive the current standard of care, no robotic pet.

INTERVENTIONS:
Behavioral: Robotic Joy for All™ pet — Patients will be provided with the robotic pet within 48 hours of admission and have access to the pets throughout their hospitalization to provide comfort and engagement.
  Arms: Robotic Pet

SUMMARY:
Robotic pets can provide a source of affection and companionship for patients. This is especially important as individuals with dementia may receive infrequent visitation from family members if their families struggle with how to cope and communicate with their loved one. Several options such as the "Joy for All™" and "Paro" robotic pets offer a source of companionship that is both interactive and comforting.

Sarasota Memorial Health Care System (SMHCS) researchers are seeking to make companion pets available to patients with dementia to provide them with a supplemental enrichment experience that enhances their overall care and lowers their risk for superimposed delirium. The intervention will consist of providing a robotic pet to the patient within 48 hours of admission, which the patient will keep with them throughout their hospital stay and upon discharge. SMHCS researchers will evaluate the effects of the robotic pet interaction on patient delirium scores, as measured by the Nursing Delirium Screening Scale (Nu-DESC), length of stay, and the use of intravenous psychotropic medications, code greys, falls occurrence, restraint use, and IV dislodgement in patients with mild-to-moderate dementia. The Nu-DESC scale is a short assessment tool, estimated to take approximately 3-5 minutes to complete and is already part of standard care at SMHCS. This tool is used by nursing staff with minimal additional training and shows consistent sensitivity (85.7%) and specificity (86.8%) in detecting delirium. The NuDESC score may be positive in a patient with dementia, since some characteristics of dementia can be similar to delirium. However, patients with dementia are at higher risk for developing delirium, so the NuDESC is a helpful tool for the nurse. A score of 2 or higher is considered screening positive for delirium. For this study, the NuDESC tool will be used as a guideline to assist in the screening of delirium. The patients will have to score a 4 or less to be included in the study. Patients that are scoring >4 will be excluded. Theoretic Framework of Acceptability (TFA) is a questionnaire which will be used to assess health care provider acceptability of the companion animal. This tool is currently not in use at SMHCS, but it will be used as part of this study to assess whether health care providers accept (or reject) the robotic pets as companion animals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with:

  * Dementia indicated in the patient's chart
  * Admitted to the designated medical-surgical units at Sarasota Memorial Health Care System
  * Ages 65 and older
  * NuDESC score will be 0-4 during study enrollment.

Exclusion Criteria:

* Patients who are:

  * <65 years old
  * NuDESC score >4 during study enrollment
  * Patients at risk for alcohol withdrawal or substance abuse withdrawal
  * Enhanced isolation precautions (c.diff)
  * Presenting with paranoia, hallucinations, or severe agitation

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2024-01-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Assess how the use of the Joy for All™ companion pet, as compared to standard care, impacts the development or progression of acute delirium in patients with dementia in an acute care setting. | Measured at shift change (12 hours intervals), or any time a change in mental status is observed. This will be assessed from the time the "robotic pet order" is placed until discharge up to 60 days.
  Delirium, measured by the Nursing Delirium Screening (Nu-DESC) scale, will be compared between intervention group and control group. The NUDESC score ranges from 0-10.
The use of intravenous psychotropic medications. | Recorded any time intravenous psychotropic medication is administered starting from the time the "robotic pet order" is placed until patient is discharge up to 60 days.
  The use of intravenous psychotropic medications (i.e. Haldol, Ativan, etc.) in patients with dementia will be compared between groups.
Hospital length of stay. | Length of stay is measured from time of admission to time of discharge up to 60 days.
  Hospital length of stay will be evaluated between the intervention group and the control group.
The use of restraints. | Use of restraints will be recorded starting from the time the "robotic pet order" is placed until patient is discharged up to 60 days.
  The use of restraints will be compared intervention group and control group.
Occurrence of falls. | Any fall that occurs during an enrolled patient's hospital stay will be recorded starting from the time the "robotic pet order" is placed until patient is discharged up to 60 days.
  The number of falls patients have during their hospital stay will be compared between the intervention group and control group.
"Code Greys" | During the length of the patient's hospitalization, any "Code Grey" will be recorded at time of occurrence starting from the time the "robotic pet order" is placed until patient is discharged up to 60 days.
  The number of "Code Greys" called will be recorded and compared between groups.
Intravenous catheter dislodgement occurrences. | All enrolled patients will have any intravenous catheter dislodgment recorded at time of occurrence. This will be recorded starting from the time the "robotic pet order" is placed until patient is discharged, up to 60 days.
  Patient's will be monitored for intravenous catheter dislodgements.
Delirium order set. | Delirium and worsening of condition will be recorded at time of observation during hospitalization stay up to 60 days.
  Any worsening of condition, evidence of delirium, or delirium order set will be monitored and recorded.
Use of patient safety attendants (order and length of use) | Patient safety attendant use and camera use will be recorded for use and length of time for each patient enrolled in the study starting from the time the "robotic pet order" is placed until patient is discharged up to 60 days.
  The group receiving the Joy for All companion pet use of patient safety attendants and/or use of cameras will be compared to the controls group use of patient safety attendants and/or cameras. Number of uses and time of use will be recorded.
Blood Pressure | Blood pressure measurements will be collected and monitored during the time the patient is admitted following standard of care procedure, from the time the "robotic pet order", and continue until patient is discharge, up to 60 days.
  Assess how the use of the Joy for All™ companion pet, as compared to standard care, impacts systolic and diastolic blood pressure in patients with mild-to-moderate dementia in an acute care setting.
Heart Rate | Heart rate measurements will be collected and monitored during the time the patient is admitted following standard of care procedure, from the time the "robotic pet order" is placed, and continue until patient is discharge, up to 60 days.
  Assess how the use of the Joy for All™ companion pet, as compared to standard care, impacts heart rates in patients with mild-to-moderate dementia in an acute care setting
Pain Signs | Signs of pain will be collected and monitored during the time the patient is admitted following standard of care procedure, from the time the "robotic pet order" is placed, and continue until patient is discharge, up to 60 days.
  Assess how the use of the Joy for All™ companion pet, as compared to standard care, impacts pain signs in patients with mild-to-moderate dementia in an acute care setting, using a 0-10 Likert scale for pain assessment.

SECONDARY OUTCOMES:
Determine the registered nurses acceptability of the Joy for All™ companion pet as a form of complementary therapy for patients with dementia in the acute setting. | Flyers will be provided to nurse leadership, charge nurses and in unit common areas (e.g., breakroom) 1-2 times a month for them to take the survey. Emails will also be sent out with the link to take the survey up to 2 years..
  Registered nurses will report Joy for All™ companion pets as an acceptable form of complementary therapy for patients with dementia as measured by the Theoretic Framework of Acceptability (TFA) Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Joanna D'Elia, MSN, RN, GERO-BC, Principal Investigator — Sarasota Memorial Health Care System
Locations (1):
- Sarasota Memorial Health Care System, Sarasota, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heidenreich, A. & Gresbach, S. (2018). The "Nu" way for nurses to screen for delirium. American Nurse Today, 13(5). 52-54.
- [Background] Hudson J, Ungar R, Albright L, Tkatch R, Schaeffer J, Wicker ER. Robotic Pet Use Among Community-Dwelling Older Adults. J Gerontol B Psychol Sci Soc Sci. 2020 Oct 16;75(9):2018-2028. doi: 10.1093/geronb/gbaa119. PMID 32789476
- [Background] Morandi A, Bellelli G. Delirium superimposed on dementia. Eur Geriatr Med. 2020 Feb;11(1):53-62. doi: 10.1007/s41999-019-00261-6. Epub 2019 Nov 14. PMID 32297232
- [Background] Morley JE. Dementia-related agitation. J Am Med Dir Assoc. 2011 Nov;12(9):611-612.e2. doi: 10.1016/j.jamda.2011.08.008. Epub 2011 Oct 5. No abstract available. PMID 21975343
- [Background] Moyle W, Bramble M, Jones C, Murfield J. Care staff perceptions of a social robot called Paro and a look-alike Plush Toy: a descriptive qualitative approach. Aging Ment Health. 2018 Mar;22(3):330-335. doi: 10.1080/13607863.2016.1262820. Epub 2016 Dec 14. PMID 27967207
- [Background] Moyle W, Bramble M, Jones CJ, Murfield JE. "She Had a Smile on Her Face as Wide as the Great Australian Bite": A Qualitative Examination of Family Perceptions of a Therapeutic Robot and a Plush Toy. Gerontologist. 2019 Jan 9;59(1):177-185. doi: 10.1093/geront/gnx180. PMID 29165558
- [Background] Moyle W, Murfield J, Jones C, Beattie E, Draper B, Ownsworth T. Can lifelike baby dolls reduce symptoms of anxiety, agitation, or aggression for people with dementia in long-term care? Findings from a pilot randomised controlled trial. Aging Ment Health. 2019 Oct;23(10):1442-1450. doi: 10.1080/13607863.2018.1498447. Epub 2018 Nov 24. PMID 30474401
- [Background] Petersen S, Houston S, Qin H, Tague C, Studley J. The Utilization of Robotic Pets in Dementia Care. J Alzheimers Dis. 2017;55(2):569-574. doi: 10.3233/JAD-160703. PMID 27716673
- See also: Delirium: when to be worried about confusion and what to do next: Update for nurses on timely assessment of this common condition in acute settings and long-term care, and why it should be treated as a medical emergency. Nursing Older People, 35(2), 6-8. — https://doi.org/10.7748/nop.35.2.6.s2
- See also: The interface between delirium and dementia in elderly adults. The Lancet Neurology, 14(8), 823-832. — https://doi.org/10.1016/S1474-4422(15)00101-5
- See also: PARO Therapeutic Robot — http://www.parorobots.com/
- See also: Delirium. [Updated 2022 Nov 19]. — https://www.ncbi.nlm.nih.gov/books/NBK470399/